CLINICAL TRIAL: NCT01011556
Title: A Phase 2 Study for Transdermal Application of Teriparatide
Brief Title: A Study for the Transdermal Application of Teriparatide
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: TransPharma Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 12641; I2Y-MC-GHFA(c) (Other: Eli Lilly and Company)
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2012-10-23 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-09

CONDITIONS: Osteoporosis
Keywords: Age Related Osteoporosis; Senile Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Parathyroid Hormone; Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 20 mcg Subcutaneous Teriparatide (Active Comparator): Received 20 micrograms (mcg) subcutaneously once daily in an unblinded manner.
  Interventions: Drug: Subcutaneous Teriparatide
- 30 mcg Transdermal Teriparatide (Experimental): Received 30 micrograms (mcg) teriparatide transdermally via a patch applied once daily. Participants were blinded to dose level.
  Interventions: Drug: Transdermal Teriparatide
- 50 mcg Transdermal Teriparatide (Experimental): Received 50 micrograms (mcg) teriparatide transdermally via a patch applied once daily. Participants were blinded to dose level.
  Interventions: Drug: Transdermal Teriparatide
- 80 mcg Transdermal Teriparatide (Experimental): Received 80 micrograms (mcg) teriparatide transdermally via a patch applied once daily. Participants were blinded to dose level.
  Interventions: Drug: Transdermal Teriparatide

INTERVENTIONS:
Drug: Subcutaneous Teriparatide — Administered subcutaneously once daily for 12 months
  Other Names: recombinant human parathyroid hormone (rhPTH) (1-34); recombinant human teriparatide; Forteo; Forsteo; LY333334
  Arms: 20 mcg Subcutaneous Teriparatide
Drug: Transdermal Teriparatide — Administered transdermally, applied once daily for 6 hours over 12 months
  Other Names: synthetic human parathyroid hormone (shPTH) (1-34); synthetic human teriparatide
  Arms: 30 mcg Transdermal Teriparatide; 50 mcg Transdermal Teriparatide; 80 mcg Transdermal Teriparatide

SUMMARY:
The primary purpose of this study is to help answer the following research questions:

1. How teriparatide given using a skin patch (transferred through the skin using the ViaDerm Teriparatide System) compares to teriparatide injected under the skin with a needle (pen injector) affects your bone density (how solid or porous your bones are).
2. The safety of the teriparatide skin patch and any side effects that might be associated with it.

DETAILED DESCRIPTION:
Teriparatide 20 micrograms (mcg) per day is currently only available as a subcutaneous (SQ) injection and many patients with severe osteoporosis for whom anabolic therapy with teriparatide is appropriate are either unwilling or physically unable to self-inject. The purpose of this Phase 2 study is to identify a transdermal dose or doses that will be comparable to the teriparatide 20 mcg SQ dose from a pharmacodynamic (PD) and safety standpoint for use in future Phase 3 studies.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory, postmenopausal women.
* Centrally confirmed lumbar spine or femoral neck bone mineral density (BMD) T-score of less than or equal to -2.5.
* Without language barrier, cooperative, expected to return for all follow-up procedures, and have given informed consent after being informed of the risks, medications, and procedures to be used in the study.
* Able to use the pen-type injection delivery system and the ViaDerm Teriparatide System satisfactorily in the opinion of the investigator, or with the help of a family member or caregiver.
* Able to be reached by telephone for follow-up contact between visits

Exclusion Criteria:

* Abnormal laboratory values for albumin and alkaline phosphatase.
* Laboratory values outside the ranges defined in the protocol for the following: Serum calcium, intact parathyroid hormone (iPTH), 25 hydroxyvitamin D, and 24-hour urine calcium
* History of diseases other than postmenopausal osteoporosis that affect bone metabolism, such as Paget's disease, renal osteodystrophy, osteomalacia, any secondary causes of osteoporosis, hypoparathyroidism, hyperparathyroidism, and intestinal malabsorption.
* History of malignant neoplasms in the 5 years prior to randomization, with the exception of superficial basal cell carcinoma or squamous cell carcinoma of the skin that has been definitively treated. Patients with carcinoma in situ of the uterine cervix treated definitively more than 1 year prior to entry into the study may be randomized.
* Use of a pacemaker.
* Known chronic dermatological disorder, such as contact dermatitis
* History of allergy or sensitivity to tapes or adhesives
* Patients prone to bleeding with coagulopathies, such as hemophilia or thrombocytopenia.
* Patients who have an increased baseline risk of osteosarcoma, Paget's disease of the bone, or unexplained elevations of alkaline phosphatase; or prior external beam, implant radiation therapy involving the skeleton, or previous primary skeletal malignancy.
* Major fracture within the past year in the femur, tibia, humerus, or radius (with or without ulna).

Treatment with:

* calcitonins in the 2 months prior to randomization.
* oral, transdermal/patch, or injectable estrogens, progestins, estrogen analogs, estrogen agonists, estrogen antagonists, selective estrogen receptor modulators, or tibolone in the 3 months prior to randomization; treatment with intravaginal estrogens in doses higher than 0.3 mg of conjugated equine estrogen, or the equivalent, for more than 3 doses per week in the 3 months prior to randomization.
* androgens or other anabolic steroids in the 6 months prior to randomization.
* fluorides in the 2 years prior to randomization. (Previous or current use of fluoridated water or topical dental fluoride treatments are permitted.)
* oral bisphosphonates for more than 2 consecutive months in the 6 months prior to randomization; treatment with intravenous bisphosphonates in the 6 months prior to randomization; treatment with more than 1 cycle of intermittent oral bisphosphonates in the 6 months prior to randomization; or having received the last cycle of this intermittent oral regimen less than 4 weeks prior to screening.
* patients receiving intravenous zoledronic acid during the 12 months prior to randomization.
* vitamin D greater than 50,000 International Units (IU) per week or with any dose of calcitriol or vitamin D analogs or agonists in the 6 months prior to randomization.
* systemic corticosteroids in the 1 month prior to randomization or for more than 30 days in the 1 year prior to randomization. (Ophthalmic, otic, topical, orally inhaled, nasally inhaled, or intra-articular corticosteroid therapy may be used without these restrictions.)
* any other drug known to significantly affect bone metabolism in the 6 months prior to randomization.
* warfarin or other coumadin anticoagulants in the 1 month prior to randomization.
* any investigational drug in the 1 month prior to entry into the study.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2009-11; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (18):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Buenos Aires, Argentina
- Estonia (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pärnu
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tallinn
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tartu
- Hungary (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Balatonfüred
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Budapest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Debrecen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Esztergom
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Győr
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szombathely
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tatabánya
- Mexico (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Guadalajara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mexico City
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Monterrey
- Romania (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lasi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Timișoara

RESULTS

PARTICIPANT FLOW:
Groups:
- 20 Mcg Subcutaneous Teriparatide: Received 20 microgram (mcg) teriparatide subcutaneously (injected) once daily in an unblinded manner.
- 30 Mcg Transdermal Teriparatide: Received 30 mcg teriparatide transdermally via a patch applied once daily. Participants were blinded to dose level.
- 50 Mcg Transdermal Teriparatide: Received 50 mcg teriparatide transdermally via a patch applied once daily. Participants were blinded to dose level.
- 80 Mcg Transdermal Teriparatide: Received 80 mcg teriparatide transdermally via a patch applied once daily. Participants were blinded to dose level.
Period: Overall Study
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Started | 58 | 56 | 55 | 64
Received at Least 1 Dose of Study Drug | 57 | 56 | 54 | 64
Completed | 52 | 48 | 45 | 51
Not Completed | 6 | 8 | 10 | 13
Not completed — Adverse Event | 1 | 3 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 4 | 4
Not completed — Sponsor decision | 0 | 1 | 1 | 2
Not completed — Inclusion/exclusion criteria not met | 2 | 1 | 3 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide | Total
Number analyzed (Participants) | 57 | 56 | 54 | 64 | 231
Age Continuous [Mean (Standard Deviation); unit: years] | 63.9 (7.2) | 65.0 (8.3) | 67.6 (8.4) | 65.1 (7.2) | 65.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 56 | 54 | 64 | 231
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 14 | 15 | 14 | 17 | 60
  Latin American | 0 | 2 | 1 | 0 | 3
  Mexican | 7 | 6 | 5 | 6 | 24
  Not Hispanic or Latino | 33 | 32 | 32 | 40 | 137
  South American | 1 | 1 | 1 | 0 | 3
  Spaniard | 2 | 0 | 1 | 1 | 4
Region of Enrollment [Number; unit: participants]
  Estonia | 4 | 1 | 6 | 4 | 15
  Hungary | 21 | 25 | 23 | 25 | 94
  Mexico | 7 | 6 | 5 | 6 | 24
  Argentina | 17 | 17 | 16 | 18 | 68
  Romania | 8 | 7 | 4 | 11 | 30

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at 12 Months
Description: Bone mineral density (BMD) of the lumbar spine was assessed by dual energy X-ray absorptiometry (DXA). BMD values are corrected data and have been standardized across the machine types (Hologic and Lunar). Analyses were performed using ANCOVA model and least square (LS) means were adjusted for baseline BMD values as a covariate and pooled site and treatment as fixed effects.
Time Frame: Baseline, 12 Months
Population: All participants who received at least 1 dose of drug and had at least 1 baseline and post-baseline lumbar spine BMD measure. Analysis was performed using intention-to-treat (ITT) principle, last observation carried forward method and ANCOVA model.
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage change in BMD
Groups:
- 20 Mcg Subcutaneous Teriparatide: Received 20 micrograms (mcg) teriparatide subcutaneously once daily in an unblinded manner.
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 54 | 54 | 51 | 60
percentage change in BMD | 7.80 [6.867 to 8.730] | 0.63 [-0.321 to 1.578] | 0.32 [-0.657 to 1.287] | 1.63 [0.739 to 2.519]
Statistical Analysis 1: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Non-Inferiority or Equivalence — A noninferiority margin of 3.5% was used; p < 0.001, ANCOVA; Analyses were performed using ANCOVA model with the baseline value as a covariate and pooled site and treatment as fixed effects; Difference in Least Square Means = -7.17, 90% CI 2-sided [-8.489 to -5.851]
Statistical Analysis 2: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Non-Inferiority or Equivalence — A noninferiority margin of 3.5% was used; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Square Means = -7.48, 90% CI 2-sided [-8.822 to -6.144]
Statistical Analysis 3: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Non-Inferiority or Equivalence — A noninferiority margin of 3.5% was used; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Square Means = -6.17, 90% CI 2-sided [-7.448 to -4.891]

2. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density (BMD) at 6 Months
Description: Bone mineral density (BMD) of the lumbar spine was assessed by dual energy X-ray absorptiometry (DXA). BMD values are corrected data and have been standardized across the machine types (Hologic and Lunar). Analyses were performed using ANCOVA model with the baseline value as a covariate and pooled site and treatment as fixed effects.
Time Frame: Baseline, 6 Months
Population: All participants who received at least 1 dose of drug and had at least 1 baseline and post-baseline lumbar spine BMD measure. Analysis was performed using intent-to-treat principal, last observation carried forward method and ANCOVA model.
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage change in BMD
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 54 | 52 | 51 | 58
percentage change in BMD | 4.74 [3.953 to 5.537] | 0.16 [-0.661 to 0.983] | 0.88 [0.051 to 1.705] | 1.19 [0.418 to 1.957]
Statistical Analysis 1: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Square Means = -4.58, 90% CI 2-sided [-5.716 to -3.452]
Statistical Analysis 2: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Square Means = -3.87, 90% CI 2-sided [-5.006 to -2.727]
Statistical Analysis 3: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, ANCOVA; [statistical method as in outcome 1, analysis 1]; Difference in Least Square Means = -3.56, 90% CI 2-sided [-4.652 to -2.464]

3. Secondary Outcome: Time Course Change of BMD Response at the Lumbar Spine
Description: To assess the time course of the treatment, the BMD data of the lumbar spine was assessed by dual energy X-ray absorptiometry (DXA) and analyzed using a mixed model repeated measures (MMRM) method, with the repeated measure occurring at each visit (for example, 6 and 12 month). BMD values are corrected data and have been standardized across the machine types (Hologic and Lunar).
Time Frame: Baseline to 6 Months and 12 Months
Population: All participants who received at least 1 dose of drug, had at least 1 baseline and post-baseline lumbar spine BMD measure. Analysis was performed using ITT principal.
Measure: Least Squares Mean (90% Confidence Interval); unit: percentage change in BMD
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 57 | 56 | 54 | 63
percentage change in BMD
  6 months (n=54, 52, 51, 58) | 4.72 [3.927 to 5.516] | 0.19 [-0.630 to 1.019] | 0.78 [-0.050 to 1.606] | 1.19 [0.421 to 1.965]
  12 months (n=52, 48, 45, 50) | 8.12 [7.181 to 9.060] | 0.62 [-0.367 to 1.601] | 0.66 [-0.348 to 1.663] | 1.93 [0.989 to 2.881]
Statistical Analysis 1: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value is for change in BMD at 6 months; MMRM Model: Percentage change in BMD = treatment+baseline+pooled site+visit+treatment*visit interaction. Repeat measure occurred at each visit; Difference in Least Square Means = -4.53, 90% CI 2-sided [-5.663 to -3.392], Standard Error of Mean 0.687
Statistical Analysis 2: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value is for change in BMD at 6 months; [statistical method as in outcome 3, analysis 1]; Difference in Least Square Means = -3.94, 90% CI 2-sided [-5.086 to -2.800], Standard Error of Mean 0.692
Statistical Analysis 3: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value is for change in BMD at 6 months; [statistical method as in outcome 3, analysis 1]; Difference in Least Square Means = -3.53, 90% CI 2-sided [-4.627 to -2.430], Standard Error of Mean 0.665
Statistical Analysis 4: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — p-value is for change in BMD at 12 months; [statistical method as in outcome 3, analysis 1]; Difference in Least Square Means = -7.50, 90% CI 2-sided [-8.856 to -6.151], Standard Error of Mean 0.818
Statistical Analysis 5: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — p-value for change in BMD at 12 months; [statistical method as in outcome 3, analysis 1]; Difference in Least Square Means = -7.46, 90% CI 2-sided [-8.835 to -6.091], Standard Error of Mean 0.830
Statistical Analysis 6: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis — p-value is for change in BMD at 12 months; [statistical method as in outcome 3, analysis 1]; Difference in Least Square Means = -6.19, 90% CI 2-sided [-7.510 to -4.860], Standard Error of Mean 0.802

4. Secondary Outcome: Percent Change From Baseline in Procollagen Type 1 N-Terminal Propeptide (P1NP)
Description: Procollagen Type 1 N-Terminal Propeptide (P1NP) is a marker of bone formation.
Time Frame: Baseline, 1 Month, 3 Months, 6 Months, 12 Months
Population: All randomized participants who received at least one dose of study drug. The intent-to-treat principle was applied.
Measure: Mean (Standard Deviation); unit: percentage change in P1NP
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 52 | 53 | 51 | 62
percentage change in P1NP
  1 month (n=49, 53, 49, 60) | 112.47 (65.390) | 19.29 (35.274) | 27.78 (31.064) | 42.06 (53.000)
  3 months (n=50, 51, 49, 59) | 174.88 (118.745) | 35.68 (50.358) | 53.53 (64.625) | 116.34 (117.697)
  6 months (n=48, 49, 48, 56) | 284.89 (228.773) | 62.99 (78.579) | 93.82 (93.575) | 221.28 (233.297)
  12 months (n=47, 46, 43, 49) | 232.41 (176.557) | 72.17 (86.747) | 97.14 (98.007) | 178.02 (181.361)
Statistical Analysis 1: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 1 month
Statistical Analysis 2: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 1 month
Statistical Analysis 3: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 1 month
Statistical Analysis 4: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 3 months
Statistical Analysis 5: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 3 months
Statistical Analysis 6: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.003, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 3 months
Statistical Analysis 7: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 6 months
Statistical Analysis 8: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 6 months
Statistical Analysis 9: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.029, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 6 months
Statistical Analysis 10: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 12 months
Statistical Analysis 11: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 12 months
Statistical Analysis 12: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.047, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 12 months

5. Secondary Outcome: Percent Change From Baseline of C-Terminal Telopeptide (CTX)
Description: C-terminal telopeptide is a marker of bone resorption.
Time Frame: Baseline, 1 Month, 3 Months, 6 Months, 12 Months
Population: All randomized participants who received at least one dose of study drug. The intent-to-treat principle was applied.
Measure: Mean (Standard Deviation); unit: percentage change in CTX
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 52 | 53 | 51 | 62
percentage change in CTX
  1 month (n=49, 53, 49, 60) | 20.57 (64.980) | 8.05 (26.070) | 13.35 (29.384) | 21.66 (46.572)
  3 months (n=50, 51, 49, 59) | 87.78 (96.777) | 30.66 (42.048) | 42.40 (58.620) | 90.36 (103.367)
  6 months (n=48, 49, 48, 56) | 123.36 (128.832) | 37.36 (52.875) | 68.63 (71.059) | 127.81 (152.725)
  12 months (n=47, 46, 43, 49) | 97.52 (109.981) | 37.75 (58.035) | 61.25 (60.862) | 114.11 (157.485)
Statistical Analysis 1: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.822, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 1 month
Statistical Analysis 2: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.406, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 1 month
Statistical Analysis 3: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.312, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 1 month
Statistical Analysis 4: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 3 months
Statistical Analysis 5: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 3 months
Statistical Analysis 6: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.952, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 3 months
Statistical Analysis 7: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 6 months
Statistical Analysis 8: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.011, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 6 months
Statistical Analysis 9: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.997, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 6 months
Statistical Analysis 10: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.003, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 12 months
Statistical Analysis 11: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.112, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 12 months
Statistical Analysis 12: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p = 0.988, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 12 months

6. Secondary Outcome: Percent Change From Baseline in Serum Procollagen Type 1 C-Propeptide (P1CP) at 1 Month
Description: Procollagen Type 1 N-Terminal Propeptide (P1NP) is a marker of bone formation.
Time Frame: Baseline, 1 Month
Population: All randomized participants who received at least one dose of study drug. The intent-to-treat principle was applied.
Measure: Median (Standard Deviation); unit: percentage change in P1CP
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 49 | 53 | 48 | 59
percentage change in P1CP | 80.10 (85.421) | 4.63 (29.694) | 12.30 (30.153) | 23.84 (44.813)
Statistical Analysis 1: Comparison: 20 Mcg Subcutaneous Teriparatide vs 30 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 1 month
Statistical Analysis 2: Comparison: 20 Mcg Subcutaneous Teriparatide vs 50 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 1 month
Statistical Analysis 3: Comparison: 20 Mcg Subcutaneous Teriparatide vs 80 Mcg Transdermal Teriparatide; Test type: Superiority or Other; p < 0.001, Wilcoxon Rank Sum Test; Pairwise comparison p-value at 1 month

7. Secondary Outcome: Convenience/Ease of Use Questionnaire (CEUQ)
Description: CEUQ consists of 5 sections and 16 questions using a 5-point Likert scale designed to collect measures for ease of use (S1), convenience of use (S2), confidence of use (S3), fear of use (S4), and overall satisfaction with therapy (S5). CEUQ is not a validated instrument.
Time Frame: baseline up to 12 months
Population: All randomized participants who received at least 1 dose of study drug and had CEUQ assessment. Last observation was carried forward, unless the last observation was also the first completed questionnaire.
Measure: Number; unit: participants
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 55 | 54 | 51 | 62
participants
  S1-Stronly Disagree | 0 | 0 | 0 | 0
  S1-Somewhat Disagree | 0 | 0 | 0 | 0
  S1-Neutral | 0 | 0 | 1 | 0
  S1-Somewhat Agree | 11 | 9 | 8 | 10
  S1-Strongly Agree | 44 | 45 | 42 | 52
  S2-Strongly Disagree | 0 | 0 | 0 | 0
  S2-Somewhat Disagree | 0 | 0 | 0 | 0
  S2-Neutral | 1 | 1 | 1 | 0
  S2-Somewhat Agree | 11 | 12 | 9 | 12
  S2-Strongly Agree | 43 | 41 | 41 | 50
  S3-Not Confident | 0 | 0 | 1 | 0
  S3-Somewhat Not Confident | 0 | 1 | 0 | 1
  S3-Neutral | 0 | 0 | 3 | 4
  S3-Somewhat Confident | 13 | 15 | 11 | 17
  S3-Very Confident | 42 | 38 | 36 | 40
  S4-Extremely Fearful | 0 | 0 | 1 | 0
  S4-Somewhat Fearful | 1 | 1 | 0 | 1
  S4-Neutral | 1 | 0 | 1 | 0
  S4-Somewhat Not Fearful | 9 | 16 | 9 | 13
  S4-Not Fearful | 44 | 37 | 40 | 48
  S5-Very Dissatisfied | 0 | 0 | 0 | 0
  S5-Somewhat Dissatisfied | 0 | 1 | 1 | 0
  S5-Neutral | 1 | 0 | 2 | 1
  S5-Somewhat Satisfied | 10 | 13 | 10 | 18
  S5-Very Satisfied | 44 | 40 | 38 | 43

8. Secondary Outcome: Change in Serum Calcium With and Without Adjustments for Serum Albumin From Predose to After 4 and 6 Hours
Description: Serum calcium adjusted for serum albumin levels is calculated using the following formula: Total Calcium + [(40 - albumin) x 0.02]. Analysis for serum calcium and albumin adjusted serum calcium were collected at predose, 4 hours (h) post-dose (PD) and 6 h PD at baseline and 12 months (mon).
Time Frame: Baseline, 12 Months
Population: All randomized participants who received at least 1 dose of study drug and had serum calcium measurements or adjusted serum calcium measurements at the indicated timepoint.
Measure: Mean (Standard Deviation); unit: millimole/Liter (mmol/L)
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 57 | 56 | 54 | 64
millimole/Liter (mmol/L)
  Baseline- predose; no adjustment (n=54,53,51,62) | 2.391 (0.0776) | 2.362 (0.0933) | 2.389 (0.0921) | 2.392 (0.0915)
  Baseline- 4 h PD; no adjustment (n=55,53,51,63) | 2.432 (0.1191) | 2.358 (0.1315) | 2.403 (0.1160) | 2.393 (0.1113)
  Baseline- 6 h PD; no adjustment (n=52,51,48,59) | 2.440 (0.1159) | 2.369 (0.0789) | 2.400 (0.1167) | 2.397 (0.1048)
  12 mon-predose; no adjustment (n=52,47,45,50) | 2.463 (0.1243) | 2.427 (0.0977) | 2.427 (0.0842) | 2.432 (0.0937)
  12 mon-4 h PD; no adjustment (n=51,46,44,51) | 2.516 (0.1815) | 2.428 (0.1024) | 2.430 (0.1199) | 2.464 (0.1042)
  12 mon-6 h PD; no adjustment (n=50,45,44,51) | 2.532 (0.1429) | 2.426 (0.0866) | 2.443 (0.0997) | 2.467 (0.0959)
  baseline-predose albumin adjusted (n=53,53,50,60) | 2.363 (0.0811) | 2.341 (0.0949) | 2.376 (0.0807) | 2.373 (0.0809)
  baseline-4 h PD; albumin adjusted (n=52,52,50,61) | 2.418 (0.1099) | 2.348 (0.1283) | 2.403 (0.0928) | 2.386 (0.1045)
  baseline-6 h PD; albumin adjusted (n=49,50,47,57) | 2.423 (0.1100) | 2.363 (0.0727) | 2.404 (0.0908) | 2.394 (0.0934)
  12 mon- predose albumin adjusted (n=52,47,45,50) | 2.461 (0.0998) | 2.432 (0.0806) | 2.449 (0.0861) | 2.442 (0.0840)
  12 mon- 4 h PD; albumin adjusted (n=51,46,44,51) | 2.523 (0.1680) | 2.438 (0.1022) | 2.458 (0.1012) | 2.482 (0.0962)
  12 mon-6 h PD; albumin adjusted (n=52,47,45,50) | 2.547 (0.1236) | 2.443 (0.0838) | 2.481 (0.1044) | 2.483 (0.1348)

9. Secondary Outcome: Change From Baseline in Urine Calcium Excretion at 6 and 12 Months
Time Frame: Baseline, 6 Months, 12 Months
Population: All randomized participants who received at least 1 dose of study drug and had urine calcium measurements at the indicated timepoint.
Measure: Mean (Standard Deviation); unit: millimole/day (mmol/day)
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 57 | 56 | 54 | 64
millimole/day (mmol/day)
  Baseline | 4.45 (1.851) | 4.21 (1.766) | 4.26 (1.673) | 4.24 (1.876)
  6 months (n=54, 50, 49, 56) | 2.02 (4.122) | 0.70 (3.467) | 1.20 (2.768) | 1.35 (2.360)
  12 months (n=51, 47, 41, 51) | 5.25 (3.694) | 4.97 (2.192) | 4.80 (2.738) | 4.51 (2.770)

10. Secondary Outcome: Change From Pre-dose and Postdose Supine and Standing SBP and DBP at Baseline (BL) and 12 Months (Mon)
Description: Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) measured at pre-dose and 30 minutes (min) and 2 hours (hr) post-dose in both the supine and standing position.
Time Frame: Pre-Dose, 30 minutes, 2 hours Post-Dose at Baseline and 12 Months
Population: All randomized participants who received at least 1 dose of study drug and had predose and postdose blood pressure measurements at the indicated timepoint and body position.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 57 | 56 | 54 | 64
mmHg
  BL, supine, SBP, 30 min (n=56,54,51,62) | -0.6 (10.71) | 2.0 (10.25) | -1.0 (11.59) | -0.8 (10.77)
  BL, supine, SBP, 2 h (n=56,56,53,63) | -0.3 (13.06) | -0.9 (10.97) | -3.5 (9.97) | -0.6 (12.91)
  BL, supine, DBP, 30 min (n=56,54,51,62) | -1.9 (7.63) | 1.4 (7.59) | -2.5 (7.50) | -1.1 (7.17)
  BL, supine, DBP, 2 h (n=56,56,53,63) | -2.1 (7.59) | -0.8 (8.51) | -3.6 (7.02) | -1.6 (7.67)
  12mon, supine, SBP, 30min (n=51,47,44,51) | 0.8 (8.52) | -2.2 (7.47) | -1.1 (8.87) | -2.0 (9.82)
  12mon, supine, SBP, 2 h (n=51,47,44,51) | -0.2 (10.71) | -1.8 (11.19) | -2.5 (9.54) | -1.9 (10.87)
  12mon, supine, DBP, 30min (n=52,48,45,51) | -1.8 (7.14) | -1.8 (6.08) | -2.1 (6.77) | -1.2 (7.25)
  12mon, supine, DBP, 2 h (n=51,47,44,51) | -1.3 (6.94) | -3.3 (7.79) | -1.3 (6.79) | -2.0 (8.59)
  BL, standing, SBP, 30 min (n=56,54,51,62) | -1.3 (9.38) | 2.5 (8.93) | -0.6 (10.65) | -0.5 (10.04)
  BL, standing, SBP, 2 h (n=56,56,53,64) | -1.7 (11.57) | -1.6 (11.03) | -3.8 (10.96) | 0.0 (12.11)
  BL, standing, DBP, 30 min (n=56,54,51,62) | -2.3 (6.56) | 0.2 (8.18) | -1.2 (8.34) | -1.2 (7.80)
  BL, standing, DBP, 2 h (n=56,56,53,64) | -2.3 (7.55) | -2.1 (7.80) | -1.1 (7.25) | -1.7 (8.84)
  12mon, standing, SBP, 30min(n=51,47,44,51) | -0.6 (10.55) | -0.9 (8.41) | 0.5 (8.68) | -0.8 (8.72)
  12mon, standing, SBP, 2 h (n=51,47,44,51) | -0.1 (11.86) | -0.4 (7.64) | -1.3 (12.97) | -0.9 (10.24)
  12mon, standing, DBP, 30 min(n=51,47,44,51 | -1.8 (7.12) | -2.4 (6.04) | -3.5 (8.09) | 1.4 (7.75)
  12mon, standing, DBP, 2 h (n=51,47,44,51) | 1.1 (6.93) | -2.0 (7.35) | -1.9 (7.70) | 0.1 (7.44)

11. Secondary Outcome: Change From Pre-dose to Postdose in Supine and Standing Heart Rate at Baseline (BL) and 12 Months (Mon).
Time Frame: Pre-dose, 30 minutes, 2 hours at Baseline and 12 Months
Population: All randomized participants who received at least 1 dose of study drug and had predose and postdose heart rate measurements at the indicated timepoint and body position.
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Groups:
- 20 Mcg Subcutaneous Teriparatide: Received 20 mcg teriparatide subcutaneously once daily in an unblinded manner.
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 57 | 56 | 54 | 64
beats per minute (bpm)
  BL, supine, 30 min (n=56,54,51,62) | 1.8 (5.66) | 1.7 (5.96) | -0.8 (7.21) | -0.6 (6.50)
  BL, supine, 2 h (n=56,56,53,63) | 1.5 (8.01) | 0.9 (5.61) | -0.8 (8.49) | -0.4 (6.90)
  BL, standing, 30 min (n=56,54,51,62) | 1.6 (6.41) | -1.0 (7.36) | 0.7 (6.68) | -1.2 (7.61)
  BL, standing, 2 h (n=56,56,53,64) | 1.0 (8.03) | -0.8 (8.51) | 0.5 (6.51) | -1.0 (8.05)
  12 mon, supine, 30 min (n=51,47,44,51) | 2.5 (4.81) | 1.4 (4.74) | -0.1 (4.06) | -0.2 (5.22)
  12 mon, supine, 2 h (n=51,47,44,51) | 1.6 (6.74) | 1.1 (6.60) | -0.3 (5.43) | -0.8 (6.69)
  12 mon, standing, 30 min (n=51,47,44,51) | 1.2 (7.35) | 0.0 (5.28) | -0.7 (5.97) | -0.4 (6.90)
  12 mon, standing, 2 h (n=51,47,44,51) | 0.9 (9.03) | 0.1 (7.36) | -0.4 (7.03) | -0.7 (7.72)

12. Secondary Outcome: Number of Participants With Parathyroid Hormone (PTH) Specific Antibody Levels
Description: Participants were tested for anti-recombinant teriparatide and anti-synthetic teriparatide titers. Either none were detected (ND) or antibodies were determined to be present if the teriparatide specific antibody titers were at least 1:8 (titer 1:8).
Time Frame: Baseline and 1, 3, 12, and 13 Months (mon)
Population: All randomized participants who received at least one dose of study drug and had antibody results.
Measure: Number; unit: participants
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 57 | 56 | 54 | 64
participants
  Baseline: anti-recombinant ND (n=57, 54, 53, 64) | 57 | 54 | 52 | 64
  Baseline:anti-recombinant titer 1:8(n=57,54,53,64) | 0 | 0 | 1 | 0
  1 mon:anti-recombinant ND (n=54,54,51,62) | 54 | 54 | 51 | 62
  1 mon:anti-recombinant titer 1:8 (n=54,54,51,62 | 0 | 0 | 0 | 0
  3 mon:anti-recombinant ND (n=55,52,51,61) | 55 | 52 | 50 | 61
  3 mon:anti-recombinant titer 1:8 (n=55,52,51,6 | 0 | 0 | 1 | 0
  12 mon:anti-recombinant ND (n=52,48,45,51) | 52 | 48 | 44 | 51
  12 mon:anti-recombinant titer 1:8 (n=52,48,45,51) | 0 | 0 | 1 | 0
  13 mon:anti-recombinant ND (n=50,46,44,50) | 50 | 46 | 43 | 50
  13 mon:anti-recombinant titer 1:8 (n=50,46,44,50) | 0 | 0 | 1 | 0
  Baseline:anti-synthetic ND (n=57,54,53,64) | 57 | 54 | 52 | 64
  Baseline:anti-synthetic titer 1:8 (n=57,54,53,64) | 0 | 0 | 1 | 0
  1 mon:anti-synthetic ND (N=54,54,51,62) | 54 | 54 | 50 | 62
  1 mon:anti-synthetic titer 1:8 (N=54,54,51,62) | 0 | 0 | 1 | 0
  3 mon:anti-synthetic ND (n=55,52,51,61) | 55 | 52 | 50 | 61
  3 mon:anti-synthetic titer 1:8 (n=55,52,51,61) | 0 | 0 | 1 | 0
  12 mon:anti-synthetic ND (n=52,48,45,51) | 52 | 48 | 44 | 51
  12 mon:anti-synthetic titer 18 (n=52,48,45,51) | 0 | 0 | 1 | 0
  13 mon:anti-synthetic ND (n=50,46,44,50) | 50 | 46 | 43 | 50
  13 mon:anti-synthetic titer 1:8 (n=50,46,44,50) | 0 | 0 | 1 | 0

13. Secondary Outcome: Pharmacokinetics Parameters: Area Under the Curve (AUC)
Description: Due to high intra-subject variability, data was not analyzed for this outcome measure.
Time Frame: Baseline, 1 Month, 3 Months, and 12 Months
Population: Due to high intra-subject variability, zero participants were analyzed on this outcome measure.
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Pharmacokinetics Parameters: Maximal Concentration (Cmax)
Description: Due to high intra-subject variability, data was not analyzed for this outcome measure.
Time Frame: Baseline, 1 Month, 3 Months, 12 Months
Population: Due to high intra-subject variability, zero participants were analyzed for this outcome measure.
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 0 | 0 | 0 | 0

15. Secondary Outcome: DRAIZE Edema Assessment at Baseline Through 13 Month Follow-up
Description: Severity of edema was categorized based on a 5 point scale: 0=no edema, 4=severe edema (defined as an area raised more than 1 millimeter and extending beyond area of exposure)
Time Frame: 13 Month follow-up
Population: All randomized participants who received at least 1 dose of study drug and had edema measurements at 13 months.
Measure: Number; unit: participants
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 41 | 39 | 39 | 43
participants
  0=no edema | 41 | 39 | 39 | 43
  1=very slight edema to 4=severe edema | 0 | 0 | 0 | 0

16. Secondary Outcome: DRAIZE Erythema Assessment at Baseline Through 13 Month Follow-up
Description: Severity of erythema was categorized based on a 5 point scale: 0=no erythema, 4=severe erythema (defined as beet red to eschar)
Time Frame: 13 Month follow-up
Population: All randomized participants who received at least 1 dose of study drug and had erythema measurements at 13 months.
Measure: Number; unit: participants
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Number analyzed (Participants) | 41 | 39 | 39 | 43
participants
  0=no erythema | 41 | 39 | 39 | 43
  1=very slight erythema to 4=severe erythema | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | 20 Mcg Subcutaneous Teriparatide | 30 Mcg Transdermal Teriparatide | 50 Mcg Transdermal Teriparatide | 80 Mcg Transdermal Teriparatide
Serious Adverse Events (participants affected / at risk) | 2/57 | 2/56 | 1/54 | 5/64
Other Adverse Events (participants affected / at risk) | 30/57 | 33/56 | 30/54 | 39/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 Mcg Subcutaneous Teriparatide (N=57) | 30 Mcg Transdermal Teriparatide (N=56) | 50 Mcg Transdermal Teriparatide (N=54) | 80 Mcg Transdermal Teriparatide (N=64)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colonic polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lobar pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20 Mcg Subcutaneous Teriparatide (N=57) | 30 Mcg Transdermal Teriparatide (N=56) | 50 Mcg Transdermal Teriparatide (N=54) | 80 Mcg Transdermal Teriparatide (N=64)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (2) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 4 (5)
Application site discolouration (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Bronchitis (Infections and infestations) | 3 (4) | 1 (1) | 1 (1) | 2 (2)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Influenza (Infections and infestations) | 3 (3) | 3 (3) | 1 (1) | 5 (5)
Nasopharyngitis (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Viral infection (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 3 (4) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 1 (1) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 1 (2) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (2) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Depression (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Hypercalciuria (Renal and urinary disorders) | 2 (2) | 1 (1) | 5 (5) | 6 (6)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (4)
Intra-abdominal haematoma (Vascular disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days